# **Informed Consent Form**

Effects of Developmental Gymnastics Exercise Program on Preschoolers' Motor Skills: A Randomized Controlled Trial

June, 10, 2020.

#### **Informed Consent Form**

Study Title: Effects of Developmental Gymnastics Exercise Program on Preschoolers' Motor Skills: A Randomized Controlled Trial

Principal Investigator: Dragan Marinković

**Introduction:** Your child is being invited to participate in a clinical trial evaluating the effects of a Developmental Gymnastics (DG) exercise program on preschoolers' motor skills. Before you decide whether your child will participate, it is important for you to understand the purpose of the study, its procedures, potential risks and benefits, and your child's rights as a participant. Please take your time to read this form carefully. You are encouraged to ask any questions you may have before deciding whether to allow your child to participate.

**Purpose of the Study:** The purpose of this study is to investigate if participation in a DG exercise program could improve gross motor skills (GMS) among preschool children compared to those in a group that attended extracurricular physical activities in a kindergarten.

### **Study Procedures:**

- Your child's motor competence will be assessed using the Test of Gross Motor Development-2 (TGMD-2) by examiners trained in physical education with prior experience in TGMD-2 measurements.
- The assessments will be conducted according to the detailed instruction manual.

#### **Potential Risks:**

- There are minimal risks associated with participation in the study, such as minor injuries or discomfort during physical activities.
- Every effort will be made to minimize these risks, and trained instructors will supervise all activities.

#### **Potential Benefits:**

- Participation in the DG exercise program may improve your child's gross motor skills, coordination, balance, and overall physical fitness.
- Your child's participation will contribute to advancing scientific knowledge in the field of early childhood motor development.

### **Confidentiality:**

- Your child's personal information will be kept confidential and only accessible to authorized study personnel.
- Data collected during the study will be used for research purposes only and will be securely stored.

# **Voluntary Participation:**

- Participation in the study is voluntary, and you have the right to refuse to allow your child to participate or to withdraw your child from the study at any time without penalty or loss of benefits.
- If you choose to withdraw your child from the study, any data collected up to that point will be kept confidential and will not be used in the analysis.

**Parent/Guardian Signature:** I have read and understood the information provided in this consent form. I have had the opportunity to ask questions, and any questions I had were answered satisfactorily. I voluntarily consent to allow my child to participate in this clinical trial.

| Parent/Guardian's Name: |
|----------------------------------------|
| Parent/Guardian's Signature: |
| Date: |
| Investigator's Signature: |
| investigator s Signature. |
| Investigator's Name: Dragan Marinković |